CLINICAL TRIAL: NCT00002719
Title: RANDOMIZED PHASE III STUDY TO EVALUATE THE VALUE OF rHuG-CSF IN INDUCTION AND OF AN ORAL SCHEDULE AS CONSOLIDATION TREATMENT IN ELDERLY PATIENTS WITH ACUTE MYELOGENOUS LEUMEKIA (AML-13 PROTOCOL)
Brief Title: Combination Chemotherapy With or Without G-CSF in Treating Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-06954; EORTC-06954; ITA-GIMEMA-AML13
Record Dates: First submitted 1999-11-01; First posted 2004-04-29 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Leukemia; Neutropenia
Keywords: untreated adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); secondary acute myeloid leukemia; adult acute monocytic leukemia (M5b); neutropenia; adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Neutropenia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Filgrastim; Amsacrine; Carmustine; Cytarabine; Etoposide; Idarubicin; Mitoxantrone; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: amsacrine
Drug: carmustine
Drug: cytarabine
Drug: etoposide
Drug: idarubicin
Drug: mitoxantrone hydrochloride
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Colony-stimulating factors such as G-CSF may increase the number of immune cells found in the bone marrow or peripheral blood and may help a person's immune system recover after chemotherapy and radiation therapy. Combining more than one drug and giving drugs in different ways may kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without G-CSF in treating older patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the role of granulocyte colony-stimulating factor given during and/or after remission induction with MICE (mitoxantrone/cytarabine/etoposide) in elderly patients with acute myelogenous leukemia (AML). II. Compare the complete remission (CR) rate and survival of these patients when treated with nearly equivalent doses of oral vs. intravenous mini-ICE (idarubicin/cytarabine/etoposide) as consolidation therapy given on an outpatient basis. III. Evaluate the feasibility of a second intensive consolidation regimen consisting of BAVC (carmustine/amsacrine/etoposide/cytarabine) followed by autologous stem cell support in patients under age 71 who are in CR and have good performance status.

OUTLINE: Randomized study. All patients are randomly assigned to Arms IA through ID for Induction. Patients who achieve CR and who have adequate organ function and performance status are then randomly assigned to Arm IIA or IIB for Consolidation. At selected centers, patients in CR after their first Consolidation course who are under age 71 and in very good clinical condition are treated on Regimen A (in lieu of a second Consolidation course). The following acronyms are used: AMSA Amsacrine, NSC-249992 ARA-C Cytarabine, NSC-63878 BAVC BCNU/AMSA/VP-16/ARA-C BCNU Carmustine, NSC-409962 DHAD Mitoxantrone, NSC-301739 G-CSF Granulocyte Colony-Stimulating Factor (Rhone-Poulenc Rorer) IDA Idarubicin, NSC-256439 MICE DHAD/ARA-C/VP-16 Mini-ICE IDA/ARA-C/VP-16 PBSC Peripheral Blood Stem Cells VP-16 Etoposide, NSC-141540 INDUCTION: Arm IA: 3-Drug Combination Chemotherapy. MICE. Arm IB: 3-Drug Combination Chemotherapy plus Hematologic Toxicity Attenuation. MICE; plus G-CSF. G-CSF during chemotherapy. Arm IC: 3-Drug Combination Chemotherapy plus Hematologic Toxicity Attenuation. MICE; plus G-CSF. G-CSF after chemotherapy. Arm ID: 3-Drug Combination Chemotherapy plus Hematologic Toxicity Attenuation. MICE; plus G-CSF. G-CSF during and after chemotherapy. CONSOLIDATION: Arm IIA: 3-Drug Combination Chemotherapy. Mini-ICE. Intravenous IDA/VP-16/ARA-C. Arm IIB: 3-Drug Combination Chemotherapy. Mini-ICE. Oral IDA/VP-16 + subcutaneous ARA-C. Regimen A: Stem Cell Mobilization followed by 4-Drug Combination Myeloablative Chemotherapy with Stem Cell Rescue. G-CSF; followed by BAVC; with PBSC.

PROJECTED ACCRUAL: 500 patients will be randomized for Induction, of whom an anticipated 238 patients will be randomized for Consolidation. If at interim analyses survival is shorter on Regimen A, that regimen will be closed.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute myeloblastic leukemia (AML) At least 30% blast cells in bone marrow smear Secondary AML eligible, as follows: Secondary to myelodysplastic syndrome (but not other myeloproliferative diseases) Secondary to cured Hodgkin's disease or other cured malignancy Secondary to alkylating agents or radiation for other reasons Acute promyelocytic leukemia (M3) referred to the collaborative Gruppo Italiano Malattie Ematologiche Maligne dell'Adulto-EORTC protocol (EORTC-06952) No blast crisis of chronic myeloid leukemia

PATIENT CHARACTERISTICS: Age: 61 to 80 Performance status: WHO 0-2 Life expectancy: No marked impairment from disease other than AML Hematopoietic: Not applicable Hepatic: Bilirubin less than 2 x ULN Renal: Creatinine less than 2 x ULN Cardiovascular: LVEF at least 50% No severe cardiac disease Pulmonary: No severe pulmonary disease Other: HIV seronegative (if tested) No uncontrolled infection No severe neurologic, metabolic, or psychiatric disease No other concomitant disease that precludes protocol therapy No other progressive malignant disease

PRIOR CONCURRENT THERAPY: No prior chemotherapy

Ages: 61 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 1995-12; Primary Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roel Willemze, MD, PhD, Study Chair — Leiden University Medical Center; Franco Mandelli, MD, Study Chair — Azienda Policlinico Umberto Primo
Locations (1):
- Azienda Policlinico Umberto Primo, Rome, Italy

REFERENCES:
- [Result] Thomas X, Suciu S, Rio B, Leone G, Broccia G, Fillet G, Jehn U, Feremans W, Meloni G, Vignetti M, de Witte T, Amadori S. Autologous stem cell transplantation after complete remission and first consolidation in acute myeloid leukemia patients aged 61-70 years: results of the prospective EORTC-GIMEMA AML-13 study. Haematologica. 2007 Mar;92(3):389-96. doi: 10.3324/haematol.10552. PMID 17339189
- [Result] Amadori S, Suciu S, Jehn U, Stasi R, Thomas X, Marie JP, Muus P, Lefrere F, Berneman Z, Fillet G, Denzlinger C, Willemze R, Leoni P, Leone G, Casini M, Ricciuti F, Vignetti M, Beeldens F, Mandelli F, De Witte T; EORTC/GIMEMA Leukemia Group. Use of glycosylated recombinant human G-CSF (lenograstim) during and/or after induction chemotherapy in patients 61 years of age and older with acute myeloid leukemia: final results of AML-13, a randomized phase-3 study. Blood. 2005 Jul 1;106(1):27-34. doi: 10.1182/blood-2004-09-3728. Epub 2005 Mar 10. PMID 15761020
- [Result] Jehn U, Suciu S, Thomas X, Lefrere F, Muus P, Berneman Z, Marie JP, Adamo F, Fillet G, Nobile F, Ricciuti F, Leone G, Rizzoli V, Montanaro M, Beeldens F, Fazi P, Mandelli F, Willemze R, de Witte T, Amadori S. Non-infusional vs intravenous consolidation chemotherapy in elderly patients with acute myeloid leukemia: final results of the EORTC-GIMEMA AML-13 randomized phase III trial. Leukemia. 2006 Oct;20(10):1723-30. doi: 10.1038/sj.leu.2404356. Epub 2006 Aug 17. PMID 16932345